CLINICAL TRIAL: NCT02477969
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Clinical Study Evaluating PEGylated Loxenatide Injection（PEX168）Combined With Metformin in the Treatment of Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of PEX168 in Combination Therapy Diabetes Mellitus Type 2 Patients With Metformin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEX168-302
Record Dates: First submitted 2015-05-30; First posted 2015-06-23 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — polyethylene glycol loxenatide; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PEX168(100µg) (Experimental): PEX168,100µg,Subcutaneous injection,once a week. Metformin,0.5mg, tid,oral.
  Interventions: Drug: PEX168(100µg); Drug: Metformin
- PEX168(200µg) (Experimental): PEX168,200µg,Subcutaneous injection,once a week. Metformin,0.5mg, tid,oral.
  Interventions: Drug: PEX168(200µg); Drug: Metformin
- Placebo (Placebo Comparator): Placebo,0.5ml,Subcutaneous injection,once a week. Metformin,0.5mg, tid,oral.
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: PEX168(100µg) — PEX168,100µg,Subcutaneous injection,once a week. continued for 52 weeks
  Other Names: Polyethylene Glycol Loxenatide
  Arms: PEX168(100µg)
Drug: PEX168(200µg) — PEX168,Subcutaneous injection,once a week. continued for 52 weeks
  Other Names: Polyethylene Glycol Loxenatide
  Arms: PEX168(200µg)
Drug: Placebo — 0.5ml,Subcutaneous injection,once a week.continued for 24 weeks,then followed by PEX168 100µg,qw sc. or 200µg qw sc.for 28 weeks.
  Other Names: PEGylated Loxenatide Injection Mimetics
  Arms: Placebo
Drug: Metformin — 0.5mg,oral,tid.
  Other Names: ge hua zhi

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, phase III clinical study that will enroll approximately 564 T2DM patients who before screening have inadequately controlled blood glucose （7.0%≤HbA1c≤10.5% at randomization）despite at least 8 weeks of metformin monotherapy at stable doses（≥1500 mg/day).

DETAILED DESCRIPTION:
Subjects will be randomized to receive either PEX168 100μg, 200μg or PEX 168 Dummy Injection as add-on to metformin hydrochloride. The baseline HbA1c level （HbA1c≤8.5% or HbA1c>8.5）is designed as the stratification factor based on which a dynamic randomization will be performed.

This study consists of 4 periods： Period 1：Up to 3 weeks of screening period. Period 2：A 4-week PEX168 dummy injection run-in period. Period 3：A 52-week treatment period (including a 24-week core treatment period and a 28-week extended treatment period).

Period 4: A 30-day safety follow-up period.

ELIGIBILITY:
Inclusion criteria：

1. Type 2 diabetes mellitus confirmed by the 1999 WHO criteria
2. Men or women
3. Age at signing the ICF≥18 years and ≤78 years
4. Body mass index (BMI) 20-40 Kg/m2
5. At least 8 weeks of metformin monotherapy received prior to screening
6. No glucose-lowering medications other than metformin received within the 8 weeks prior to screening
7. 7.5%≤HbA1c≤11.0% at screening（local or centralized test 7.0%≤HbA1c≤10.5% at randomization (centralized test)
8. Ability to understand the procedures and approach of this study, willingness to complete the study in strict compliance with the protocol and to voluntarily sign the ICF

Exclusion criteria (subject to be excluded if meeting any of the followings)

1. Investigator suspecting the subject of allergy to the study drug
2. Use of any of the following medications or therapies prior to screening

   * GLP-1 receptor agonists, GLP-1 analogues, DPP-4 inhibitors or any other incretin analogues
   * Growth hormone therapy within the 6 months prior to screening
   * History of drug abuse or alcohol abuse
   * Participation in any clinical trial for a pharmaceutical product or medical device within the 3 months prior to screening
   * Prolonged (for at least 7 consecutive days) intravenous, oral or intraarticular treatment with corticosteroids within the 2 months prior to screening
   * Use of any weight control agents or surgeries that might lead to unstable weight within the 2 months prior to screening, or subjects currently on a weight loss plan not in the maintenance phase
   * Any medications used prior to screening that at the investigator's discretion may confound the interpretation of the efficacy or safety data, or use of any medications that may cause common toxicities to major organs, including Chinese herbal medicine
3. History or evidence of any of the following conditions prior to screening：

   * Type 1 diabetes mellitus, single gene mutation DM, DM associated with pancreatic injury， or secondary DM, e.g., DM secondary to Cushing syndrome or acromegalia
   * History of hypertension with SBP>160 mmHg and/or DBP>100 mmHg despite glucose-lowering agents at stable dose (for at least 4 weeks)
   * History of acute/chronic pancreatitis, history of symptomatic cholecystopathy, and the risk factors for pancreatitis including pancreatic injury
   * History of myeloid C-cell carcinoma, history of multiple endocrine neoplasm （MEN） 2A or 2B syndrome, or related familiar history
   * Clinically significant gastric emptying disorders, severe chronic gastrointestinal disorders, prolonged treatment with peristalsis stimulants, or gastrointestinal surgery
   * History of severe hypoglycemic episode, or severe hypoglycemia without symptoms
   * Significant hematological disorders , or any diseases that may lead to hemolysis or unstable RBC
   * Severe diabetic complications (e.g., macrovascular and microvascular complications) that in the opinion of the investigator make the subject not suitable to participate in this study
   * Tumors of any organ or system that have or have not been treated within the 5 years prior to screening, regardless of whether there is evidence of relapse or metastasis, with the exception of local basal cell carcinoma of the skin
   * Coronary angioplasty, coronary stenting, coronary artery bypass, uncompensated heart failure （NYHA Class III or IV）, stroke or transient cerebral ischemic attack, unstable angina, myocardial infarction, and persistent and clinically significant arrhythmia, experienced within the 6 months prior to screening
   * Acute metabolic complications (e.g., ketoacidosis, lactic acidosis, hyperosmolar coma) within the 6 months prior to screening
   * Thyroid dysfunction treated with unstable therapeutic doses (e.g., thioureas, thyroid hormones) within the 6 months prior to screening
   * Blood lipid disorders treated with unstable therapeutic doses (e.g., statins, fibrates) within the 6 months prior to screening
   * Any severe trauma or severe infection that may interfere with BG control within the 1 month prior to screening
4. Laboratory indicators meeting any of the following criteria prior to screening (any test meeting the criteria must be repeated within 3 work days for confirmation)

   * ALT>2.5×ULN and/or AST>2.5×ULN and/or total bilirubin>2.5×ULN
   * Hemoglobin≤100 g/L
   * Serum creatinine>1.5×UNL and eGFR < 45 ml/min/1.73 m2 eGFR is calculated as：186.3 ×[（Serum Creatinine（mmol/L）/88.4）]-1.154 × [Age (years)]- 0.203 × 1.223 × 0.742 （Females） or ×1（Males）
   * Serum thyroid-stimulating hormone（TSH） out of the reference range that is assessed as clinically significant by the investigator
   * Fasting TGL>5.64 mmol/L（500 mg/dl)
   * Blood amylase and urine amylase>ULN that is assessed as clinically significant by the investigator
   * Any clinically significant laboratory abnormalities that at the investigator's discretion may confound the interpretation of the efficacy or safety data
5. Clinically significant 12-lead ECG abnormalities, e.g., Grade II or III atrial ventricular block （with the exception of right bundle branch block），long QT syndrome or QTc>500ms
6. Blood donation or loss≥400 mL，or receipt of blood donation within the 4 weeks prior to screening
7. Pregnant or lactating women, or men or women of child-bearing potential not willing to take contraceptive measures during the study
8. Any other conditions of the subject that at the investigator's discretion may compound the interpretation of the efficacy or safety data

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2014-02-27 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline to Week24
  HbA1c change from baseline to treatment Week 24 when receiving PEX 168 combined with metformin hydrochloride as compared to the placebo combined with metformin hydrochloride；PEX 168 as compared to the placebo, given on the basis of diet control and exercise.

SECONDARY OUTCOMES:
The proportion of HbA1c <6.5% and <7% at the end of the analysis. | Baseline to Week24
  The proportion of HbA1c <6.5% and <7% at the end of the analysis, and the proportion receiving salvage therapy.
Fasting plasma glucose | Baseline to Week52
6 points glucose of fingertip | Baseline to Week52
  Each test point of time was before breakfast, 2 hours after breakfast, before lunch,2 hours after lunch , dinner, 2 hours after dinner.This test was performed four times including baseline,V19,V31 and V59.
Postprandial blood glucose two hours | Baseline to Week52
Postprandial blood glucose two hours AUC | Baseline to Week52
Lipid | Baseline to Week52
Weight measured by standardized procedure. | Baseline to Week52
  Collect weight data in the morning of screening period, baseline,4,8,12,18,24,38,52 weeks by standardized procedure.
Blood pressure | Baseline to Week52
  Collect blood pressure data in the morning of screening period, baseline,4,8,12,18,24,38,52 weeks by standardized procedure.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Baseline to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, MD, Principal Investigator — Shanghai the sixth Hospital
Locations (1):
- Shanghai sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No